CLINICAL TRIAL: NCT00842868
Title: The CASABLANCA Study: Catheter Sampled Blood Archive in Cardiovascular Diseases. An Observational Biomarker Study
Brief Title: The CASABLANCA Study: Catheter Sampled Blood Archive in Cardiovascular Diseases
Acronym: CASABLANCA
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, James L. Januzzi, Dr., Massachusetts General Hospital
Other Study IDs: 2008P001076
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Atherosclerosis; Contrast Induced Nephropathy; Renal Impairment
Keywords: atherosclerosis; contrast induced nephropathy; renal impairment; catheterization
MeSH Terms: conditions — Atherosclerosis; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to determine the relationship between novel blood tests for heart function (including hormones and heart enzymes measured in the blood), and assess for kidney damage before and after angiography (cardiac catheterization). We hypothesize that these novel tests will enable us to predict possible complications of catheterization immediately after the procedure.

DETAILED DESCRIPTION:
The purpose of this research is to determine the relationship between (novel) cardiac and renal biomarkers before and after angiography. Clearly, having data immediately forewarning the clinician that cardiomyocyte injury has occurred, or that impending renal failure is ahead would allow for therapeutic intervention to reduce the likelihood for severe complications, and would ultimately pave the way for opportunities to derive methods to better prevent these complications. With the rapid evolution of organ-specific markers of injury comes an opportunity to explore new venues for their application.

With respect to myocardial injury, a new highly sensitive troponin molecule testing assays have recently been validated which enables to detect extremely small concentrations of troponin released in the circulation. With these assays, it may be possible to detect possible troponin release as early as minutes after injury has occurred.

Accordingly, as a primary goal of the CASABLANCA study, we will examine the release of high sensitivity troponin assays during catheterization and correlate with clinical and standard biochemical measures in order to see if a gradient of change during catheterization would be associated with subsequent recognition of peri-procedural myocardial infarction; it is the expectation that ultra high-sensitivity troponin methods will allow for nearly immediate recognition of complications following heart catheterization, when compared to the standard, non-high sensitivity methods currently in use.

With regards to peri-procedural renal injury, at present, several serum markers are being studied as potential markers or predictors in contrast induced nephropathy (CIN): Neutrophil gelatinase-associated lipocalin (NGAL) is highly accumulated in the kidney cortical tubules and leaks into the circulation after nephrotoxic and ischemic injuries. Up-regulation of the neutrophil adhesion receptor CD11b has also been associated with acute renal injury after cardiac surgery, while carbamylated hemoglobin performed quite well in differentiating acute kidney injury from elevated creatinine due to chronic kidney disease. Finally, Cystatin-C has shown to have a good accuracy for the early diagnosis of acute kidney injury before the clinical diagnosis as well.

In addition, blood will be stored for future testing of novel and experimental biomarkers in 'bench-to-bedside' collaborations, as a final yet crucial step in translational research.

ELIGIBILITY:
Inclusion Criteria:

* evaluation for possible or confirmed coronary artery disease with or without intervention
* evaluation of cerebrovascular and/or peripheral artery disease with or without intervention

Exclusion Criteria:

* Inability or unwillingness to participate
* Procedures without angiographic procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1250 patients undergoing angiography as clinical standard (diagnostic or therapeutic) care;
Sampling Method: Non-Probability Sample
Enrollment: 1298 (Actual)
Dates: Start 2008-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
major cardiovascular event | 1 year follow up

SECONDARY OUTCOMES:
renal dysfunction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James L Januzzi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bellomo TR, Liu Y, Gilliland TC, Miksenas H, Haidermota S, Wong M, Hu X, Cristino JR, Browne A, Plutzky J, Tsimikas S, Januzzi JL Jr, Natarajan P. Associations between lipoprotein(a), oxidized phospholipids, and extracoronary vascular disease. J Lipid Res. 2024 Jul;65(7):100585. doi: 10.1016/j.jlr.2024.100585. Epub 2024 Jun 26. PMID 38942114
- [Derived] Januzzi JL Jr, van Kimmenade RRJ, Liu Y, Hu X, Browne A, Plutzky J, Tsimikas S, Blankstein R, Natarajan P. Lipoprotein(a), Oxidized Phospholipids, and Progression to Symptomatic Heart Failure: The CASABLANCA Study. J Am Heart Assoc. 2024 Jun 18;13(12):e034774. doi: 10.1161/JAHA.124.034774. Epub 2024 Jun 11. PMID 38860394
- [Derived] Adusumalli S, Mohebi R, McCarthy CP, Megaret CA, Rhyne RF, Jaffer FA, Januzzi JL. Multiple Biomarkers to Predict Major Adverse Cardiovascular Events in Patients With Coronary Chronic Total Occlusions. medRxiv [Preprint]. 2023 Jul 23:2023.07.19.23292911. doi: 10.1101/2023.07.19.23292911. PMID 37503157
- [Derived] Gilliland TC, Liu Y, Mohebi R, Miksenas H, Haidermota S, Wong M, Hu X, Cristino JR, Browne A, Plutzky J, Tsimikas S, Januzzi JL Jr, Natarajan P. Lipoprotein(a), Oxidized Phospholipids, and Coronary Artery Disease Severity and Outcomes. J Am Coll Cardiol. 2023 May 9;81(18):1780-1792. doi: 10.1016/j.jacc.2023.02.050. PMID 37137588
- [Derived] Mohebi R, Murphy S, Jackson L, McCarthy C, Abboud A, Murtagh G, Gawel S, Miksenas H, Gaggin H, Januzzi JL Jr. Biomarker prognostication across Universal Definition of Heart Failure stages. ESC Heart Fail. 2022 Dec;9(6):3876-3887. doi: 10.1002/ehf2.14071. Epub 2022 Aug 8. PMID 35942508
- [Derived] Mohebi R, van Kimmenade R, McCarthy C, Gaggin H, Mehran R, Dangas G, Januzzi JL Jr. A Biomarker-Enhanced Model for Prediction of Acute Kidney Injury and Cardiovascular Risk Following Angiographic Procedures: CASABLANCA AKI Prediction Substudy. J Am Heart Assoc. 2022 May 17;11(10):e025729. doi: 10.1161/JAHA.122.025729. Epub 2022 May 16. PMID 35574956
- [Derived] Mohebi R, Jackson L, McCarthy CP, Murtagh G, Murphy SP, Abboud A, Miksenas H, Gaggin HK, Januzzi JL Jr. Relation of High-Sensitivity Cardiac Troponin I and Obstructive Coronary Artery Disease in Patients Without Acute Myocardial Infarction. Am J Cardiol. 2022 Jun 15;173:16-24. doi: 10.1016/j.amjcard.2022.03.001. Epub 2022 Mar 28. PMID 35361478
- [Derived] McCarthy CP, Shrestha S, Ibrahim N, van Kimmenade RRJ, Gaggin HK, Mukai R, Magaret C, Barnes G, Rhyne R, Garasic JM, Januzzi JL. Performance of a clinical/proteomic panel to predict obstructive peripheral artery disease in patients with and without diabetes mellitus. Open Heart. 2019 May 13;6(1):e000955. doi: 10.1136/openhrt-2018-000955. eCollection 2019. PMID 31217993
- [Derived] Natarajan P, Collier TS, Jin Z, Lyass A, Li Y, Ibrahim NE, Mukai R, McCarthy CP, Massaro JM, D'Agostino RB Sr, Gaggin HK, Bystrom C, Penn MS, Januzzi JL Jr. Association of an HDL Apolipoproteomic Score With Coronary Atherosclerosis and Cardiovascular Death. J Am Coll Cardiol. 2019 May 7;73(17):2135-2145. doi: 10.1016/j.jacc.2019.01.073. PMID 31047001
- [Derived] Elmariah S, McCarthy C, Ibrahim N, Furman D, Mukai R, Magaret C, Rhyne R, Barnes G, van Kimmenade RRJ, Januzzi JL Jr. Multiple biomarker panel to screen for severe aortic stenosis: results from the CASABLANCA study. Open Heart. 2018 Nov 1;5(2):e000916. doi: 10.1136/openhrt-2018-000916. eCollection 2018. PMID 30487984
- [Derived] McCarthy CP, Ibrahim NE, Lyass A, Li Y, Gaggin HK, Simon ML, Mukai R, Gandhi P, Kelly N, Motiwala SR, van Kimmenade RRJ, Massaro JM, D'Agostino RB Sr, Januzzi JL Jr. Single-Molecule Counting of High-Sensitivity Troponin I in Patients Referred for Diagnostic Angiography: Results From the CASABLANCA (Catheter Sampled Blood Archive in Cardiovascular Diseases) Study. J Am Heart Assoc. 2018 Mar 8;7(6):e007975. doi: 10.1161/JAHA.117.007975. PMID 29519811
- [Derived] Ibrahim NE, Lyass A, Gaggin HK, Liu Y, van Kimmenade RRJ, Motiwala SR, Kelly NP, Gandhi PU, Simon ML, Belcher AM, Harisiades JE, Massaro JM, D'Agostino RB, Januzzi JL Jr. Predicting new-onset HF in patients undergoing coronary or peripheral angiography: results from the Catheter Sampled Blood Archive in Cardiovascular Diseases (CASABLANCA) study. ESC Heart Fail. 2018 Jun;5(3):240-248. doi: 10.1002/ehf2.12268. Epub 2018 Feb 9. PMID 29424480
- [Derived] McCarthy CP, van Kimmenade RRJ, Gaggin HK, Simon ML, Ibrahim NE, Gandhi P, Kelly N, Motiwala SR, Belcher AM, Harisiades J, Magaret CA, Rhyne RF, Januzzi JL Jr. Usefulness of Multiple Biomarkers for Predicting Incident Major Adverse Cardiac Events in Patients Who Underwent Diagnostic Coronary Angiography (from the Catheter Sampled Blood Archive in Cardiovascular Diseases [CASABLANCA] Study). Am J Cardiol. 2017 Jul 1;120(1):25-32. doi: 10.1016/j.amjcard.2017.03.265. Epub 2017 Apr 12. PMID 28487034
- [Derived] Ibrahim NE, Januzzi JL Jr, Magaret CA, Gaggin HK, Rhyne RF, Gandhi PU, Kelly N, Simon ML, Motiwala SR, Belcher AM, van Kimmenade RRJ. A Clinical and Biomarker Scoring System to Predict the Presence of Obstructive Coronary Artery Disease. J Am Coll Cardiol. 2017 Mar 7;69(9):1147-1156. doi: 10.1016/j.jacc.2016.12.021. PMID 28254177
- [Derived] Gaggin HK, Liu Y, Lyass A, van Kimmenade RR, Motiwala SR, Kelly NP, Mallick A, Gandhi PU, Ibrahim NE, Simon ML, Bhardwaj A, Belcher AM, Harisiades JE, Massaro JM, D'Agostino RB Sr, Januzzi JL Jr. Incident Type 2 Myocardial Infarction in a Cohort of Patients Undergoing Coronary or Peripheral Arterial Angiography. Circulation. 2017 Jan 10;135(2):116-127. doi: 10.1161/CIRCULATIONAHA.116.023052. Epub 2016 Nov 21. PMID 27881568